CLINICAL TRIAL: NCT06635564
Title: Personalized ViscoElastic Testing-guided Bleeding Management In Liver Surgery, Neurosurgery and Obstetrics - a Prospective Comparison of the Novel ClotPro With ROTEM and TEG
Brief Title: Personalized ViscoElastic Testing-guided Bleeding Management In Liver Surgery, Neurosurgery and Obstetrics
Acronym: VETILNO
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Synapse - Research Institute Maastricht (Unknown)
Responsible Party: Principal Investigator, Johannes Gratz, Principal investigator, Medical University of Vienna
Other Study IDs: 1622/2023
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Thrombelastography; Liver Transplant; Postpartum Hemorrhage; Bleeding Disorder; Intracranial Hemorrhages
Keywords: Viscoelastic testing; personalized bleeding management
MeSH Terms: conditions — Postpartum Hemorrhage; Hemostatic Disorders; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with functional liver disease undergoing liver surgery: This group consists of patients with liver disease undergoing elective liver surgery defined as one of the following invasive procedures a) liver resection (anatomic or non-anatomic segmental resection, right or left hepatectomy, right or left extended hepatectomy) or b) orthotopic liver transplantation.
  Interventions: Diagnostic Test: Viscoelastic testing
- neurosurgical patients undergoing intracranial procedures: This group consists of patients who undergo elective neurosurgery e.g. tumor resection, aneurysm clipping or other intracranial procedures.
  Interventions: Diagnostic Test: Viscoelastic testing
- pregnant women undergoing cesarean section: This group consists of pregnant women undergoing elective cesarean section.
  Interventions: Diagnostic Test: Viscoelastic testing

INTERVENTIONS:
Diagnostic Test: Viscoelastic testing — viscoelasting testing refers to a global hemostatic assay,that quantifies the viscoelastic properties of citrated whole blood

SUMMARY:
The ClotPro analyzer is a new generation viscoelastic analyzer for the in vitro assessment of blood coagulation. This study aims to assess the agreement of ClotPro 6.0, ROTEM delta, and TEG 6s in three distinct cohorts: i) patients with liver disease undergoing liver surgery, ii) pregnant women undergoing elective cesarean section, and iii) patients undergoing elective intracranial neurosurgery. Further coagulation tests will be performed (standard laboratory coagulation tests, thrombin and plasmin generation tests) in an exploratory fashion to compare them with viscoelastic test results. The obtained test results will not result in any diagnostic or therapeutic consequences for patients included in this study.

DETAILED DESCRIPTION:
The primary research question is therefore to compare various parameters of standard ClotPro measurements with corresponding ROTEM delta and TEG 6s parameters.

Additionally, this study aims to close the following clinically important knowledge gaps:

Do VET results mirror measurements obtained by more holistic, in-depth analyses of the hemostatic system that are currently not available in clinical practice, such as TGA-TM and PG?

Which of the three investigated VET devices offers the most rapid availability of diagnostic results?

Do VET results have a predictive ability for the occurrence of perioperative bleeding and/or thromboembolic events?

Do VET results depict sex-specific differences in perioperative coagulation management?

Furthermore, by including a large number of patients from three distinct patient cohorts, this study intends to examine whether cohort-specific reference ranges need to be established for ClotPro. Thereby, this study aims to provide the foundation for an evidence-based ClotPro-guided perioperative coagulation management algorithm, which could upscale current opportunities of personalizing perioperative coagulation management.

ELIGIBILITY:
Inclusion Criteria:

1. Vulnerable patient cohorts

   * Patients undergoing elective liver surgery defined as one of the following invasive procedures:

     * Liver resection (anatomic or non-anatomic segmental resection, right or left hepatectomy, right or left extended hepatectomy),
     * Orthotopic liver transplantation,
   * Pregnant women undergoing an elective caesarean section, and
   * Patients undergoing an elective intracranial neurosurgery.
2. Written informed consent

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of three groups:
  1. Patients with liver disease undergoing elective liver surgery defined as one of the following invasive procedures a) liver resection (anatomic or non-anatomic segmental resection, right or left hepatectomy, right or left extended hepatectomy) or b) orthotopic liver transplantation.
  2. Pregnant women undergoing elective cesarean section.
  3. Patients undergoing elective intracranial neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Limits of agreement viscoelastic test parameters | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  Calculate limits of agreement between the following corresponding viscoelastic test parameters:
  * EX-test- clotting time vs. EXTEM-clotting time vs. citrated rapid TEG r time
  * EX-test- maxium clot firmness vs. EXTEM-maximum clot firmness vs. citrated rapid TEG-maximum amplitude
  * FIB-test-clotting time vs. FIBTEM-clotting time vs. citrated functional fibrinogen r time
  * FIB-test-maxium clot firmness vs. FIBTEM-maxium clot firmness vs. citrated functional fibrinogen-maximal amplitude

SECONDARY OUTCOMES:
In depth hemostatic assessment: Viscoelastic tests (VET) & thrombin generation assay (with thrombmodulin) | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  Correlation between the following viscoelastic test parameters and thrombin generation (TG) measurements:
  - Ex-test clotting time, citrated rapid TEG r time and the ratio of endogenous thrombin potential derived by TG assay using thrombomodulin
In depth hemostatic assessment: Viscoelastic tests (VET) & standard laboratory coagulation tests (SLT) | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  Correlation between the following VET parameters and SLT measurements:
  * EX-test clotting time and citrated rapid TEG r time vs. prothrombin time and
  * FIB-test maximum clot firmness, citrated functional fibrinogen-maximal amplitude and citrated functional fibrinoge- functional level of fibrinogen vs. Clauss fibrinogen.
In depth hemostatic assessment: Viscoelastic tests & plasmin generation (PG) | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  Correlation between the viscoelastic test parameters TPA-lysis time and TPA-maximal lysis with the endogenous plasmin potential derived by plasmin generation measurements.
Patient cohort-specific reference ranges | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  This anaylsis aims to investigate whether there is a need for cohort-specific reference ranges for ClotPro by assessing the distributional differences of ClotPro results between three patient cohorts (patients undergoing liver surgery, pregnant women undergoing elective cesarean section, patients undergoing an elective intracranial neurosurgery)
Useability | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  To evaluate the clinical useability of the three viscoelastic test devices by assessing differences in time from starting sample processing until each device reports the following parameters: clot formation (CT / R) and clot firmness (MCF / MA)
Predictability of clinical outcome: blood products | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  To assess wether baseline clot formation (CT / R) and clot firmness (MCF / MA) measurements for the extrinsic VET coagulation assays (EX-test, EXTEM, and CRT; FIB-test, FIBTEM, and CFF) correlate with the amount of blood product consumption.
Predictability of clinical outcomes: hemorrhage | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  To examine whether end of surgery clot formation (CT / R) and clot firmness (MCF / MA) measurements derived by viscoelastic test assays (EX-test, EXTEM, and CRT; FIB-test, FIBTEM, and CFF) correlate with hemorrhage defined by cCT imaging in patients undergoing intracranial neurosurgery.
Predictability of clinical outcomes: ocurrence of BIMS (Bleeding Independently associated with Mortality after noncardiac Surgery) or need for surgical bleeding control | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  To examine wether end of surgery clot formation (CT / R) and clot firmness (MCF / MA) measurements for the viscoelastic test assays (EX-test, EXTEM, and CRT; FIB-test, FIBTEM, and CFF) correlate with the occurrence of i) BIMS, ii) the need for interventional radiologic procedures to stop bleeding within the surgical site, or iii) the need for revision in the operating room within the first 30 postoperative days.
Predictability of clinical outcomes: thromboembolism | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24) Edit
  To examine whether a combination of baseline and end of surgery clot formation (CT / R) and clot firmness (MCF / MA) measurements for the viscelastic test assays (EX-test, EXTEM, and CRT; FIB-test, FIBTEM, and CFF) correlate with the occurrence of i) DVT (deep venous thrombosis), ii) PE (pulmonary embolism), ii) PVT (portal vein thrombosis) within the first 30 postoperative days.
Coagulational differences based on biological sex | Baseline (immediately after induction of general anaesthesia / prior to regional anesthesia); end of the surgery / intervention (assessed up to 1h); Day 1: 1. postoperative day (assessed within 24h) ; Day 3: 3. postoperative day (assessed within 24)
  In this analysis, differences in the coagulational profile as assessed by viscoelastic tests, standard laboratory coagulation tests, thrombin generation assays (with thrombomodulin) and plasmin generation measurements will be compared between subjects of female or male sex.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Gratz, PhD MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
* Study Protocol
  * Statistical Analysis Plan (SAP)
  * Informed Consent Form (ICF)
  * Clinical Study Report (CSR)
  * Analytic Code